CLINICAL TRIAL: NCT05856760
Title: A Multicentered, Single-group Phase 2, Exploratory, Open-label Study to Investigate Safety and Effect of Sparsentan in Combination With SGLT2 Inhibition in the Treatment of Adult Participants With Immunoglobulin A Nephropathy (IgAN)
Brief Title: A Study to Investigate Safety and Effect of Sparsentan in Combination With SGLT2 Inhibition in Participants With IgAN
Acronym: SPARTACUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVTX-RE021-204
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Immunoglobulin A Nephropathy
Keywords: IgAN
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — sparsentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sparsentan (Experimental): Sparsentan will be administered daily as a 200-mg oral tablet. The goal is to titrate from the initial dose of 200 mg (Day 1) to the target dose of 400 mg at Week 2.
  Interventions: Drug: Sparsentan

INTERVENTIONS:
Drug: Sparsentan — Target dose of 400 mg daily
  Other Names: Filspari; RE-021

SUMMARY:
This was a 28-week, open-label, multicenter, single-group Phase 2 exploratory study to determine the safety and effect of sparsentan in participants with IgAN who are at risk of disease progression to kidney failure despite being on both stable RAASi and SGLT2 inhibitor treatment for at least 12 weeks prior to study entry

DETAILED DESCRIPTION:
This was a 28-week, open-label, multicenter, single-group Phase 2 exploratory study to determine the safety and effect of sparsentan in participants with Immunoglobulin A Nephropathy (IgAN) who are at risk of disease progression to kidney failure (KF) despite being on both stable renin angiotensin aldosterone system inhibitor (RAASi) and sodium glucose cotransporter-2 (SGLT2) inhibitor treatment for at least 12 weeks prior to study entry.

Participants who provided written informed consent were assessed for eligibility and underwent baseline evaluations including clinical laboratory tests. Per the eligibility criteria, all participants were required to be on a stable dose(s) of angiotensin converting enzyme inhibitor (ACEI) and/or angiotensin receptor blocker (ARB) and on a stable dose of a SGLT2 inhibitor at screening and continued their stable treatments through the screening period. Eligible participants discontinued ACEI and/or ARB therapy the day before the Day 1 visit and remained on stable SGLT2 inhibitor dosing for the duration of the study.

Study intervention was administered daily for a treatment period of 24 weeks with study visits conducted at weeks 2-, 4-, 12-, and 24- following Day 1. Following the 24-week treatment period, study intervention was discontinued for 4 weeks and standard of care RAASi treatment resumed, with a safety visit at Week 28.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at the time of signing the informed consent.
* Biopsy-proven IgAN. The biopsy may have been performed at any time in the past.
* UA/C ≥0.3 g/g at screening
* An eGFR value of ≥25 mL/min/1.73m^2 at screening.
* On a stable dose of an SGLT2 inhibitor for at least 12 weeks prior to screening.
* On a stable dose of ACEI and/or ARB therapy for at least 12 weeks prior to screening that is:

  * The participant's maximum tolerated dose (MTD), and
  * at least one half of the maximum labeled dose (MLD)
* Systolic BP must be ≤160 mmHg, and diastolic BP must be ≤110 mmHg at screening.
* For participants receiving chronic low dose systemic corticosteroids (defined as ≤10 mg/day prednisone or equivalent), or an enteric formulation of budesonide and/or a mineralocorticoid receptor antagonist (MRA), the dosage must be stable for ≥12 weeks prior to screening.

Exclusion Criteria:

* IgAN secondary to another condition or immunoglobulin A (IgA) vasculitis.
* Undergone any organ transplant, with the exception of corneal transplants.
* Documented history of heart failure.
* Taking high dose (defined as >10 mg/day prednisone) or other any systemic immunosuppressive medications within 12 weeks of prior to screening.
* Has clinically significant cerebrovascular disease (transient ischemic attack or stroke) and/or coronary artery disease (hospitalization for myocardial infarction unstable angina, new onset of angina with positive functional tests, coronary angiogram revealing stenosis, or a coronary revascularization procedure) within 3 months prior to screening.
* Has jaundice, hepatitis, or known hepatobiliary disease (excluding asymptomatic cholelithiasis), or ALT and/or AST >2 times the ULN range at screening.
* Has a history of malignancy other than adequately treated basal cell or squamous cell skin cancer or cervical carcinoma within the past 2 years.
* Has a history of serious side effect or allergic response to any AngII antagonist, ERA or sparsentan, or has a hypersensitivity to any of the excipients in the study intervention.
* Requires any of the prohibited concomitant medications.
* Treatment with sparsentan within 12 weeks prior to screening
* Has participated in a study of another investigational product within 28 days prior to screening or plans to participate in such a study during the course of this study.
* Has a screening hematocrit value <27% (0.27 Volume/Volume) or hemoglobin value <9 g/dL (90 g/L).
* Has a screening potassium value of >5.5 mEq/L (5.5 mmol/L).
* Is pregnant, plans to become pregnant during the course of the study, or is breastfeeding.
* The participant, in the opinion of the Investigator, is unable to adhere to the requirements of the study, including the ability to swallow the study intervention capsules whole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Radko Komers, MD, PhD, Study Director — Travere Therapeutics, Inc.
Locations (29):
- United States (24):
  - Travere Investigational Site, Birmingham, Alabama
  - Travere Investigational Site, Chula Vista, California
  - Travere Investigational Site, Garden Grove, California
  - Travere Investigational Site, Glendale, California
  - Travere Investigational Site, Denver, Colorado
  - Travere Investigational Site, Boise, Idaho
  - Travere Investigational Site, Chubbuck, Idaho
  - Travere Investigational Site, Idaho Falls, Idaho
  - Travere Investigational Site, Chicago, Illinois
  - Travere Investigational Site, Evergreen Park, Illinois
  - Travere Investigational Site, Fort Wayne, Indiana
  - Travere Investigational Site, Kansas City, Kansas
  - Travere Investigational Site, Louisville, Kentucky
  - Travere Investigational Site, Shreveport, Louisiana
  - Travere Investigational Site, Albuquerque, New Mexico
  - Travere Investigation Site, Clifton Park, New York
  - Travere Investigational Site, Fresh Meadows, New York
  - Travere Investigational Site, New York, New York
  - Travere Investigational Site, Jacksonville, North Carolina
  - Travere Investigational Site, New Bern, North Carolina
  - Travere Investigational Site, Columbus, Ohio
  - Travere Investigational Site, Philadelphia, Pennsylvania
  - Travere Investigational Site, Columbia, South Carolina
  - Travere Investigational Site, Dallas, Texas
- Hong Kong (5):
  - Travere Investigational Site, Hong Kong
  - Travere Investigational Site, Kowloon
  - Travere Investigational Site, Shatin
  - Travere Investigational Site, Sheung Wan
  - Travere Investigational Site, Tsuen Wan

IPD SHARING:
Plan to Share IPD: Yes
Requests for clinical trial data, including language stating its intended use, should be directed to datarequest@travere.com. If approved, the requested information will be provided to the requestor after signing a data access agreement. Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication. Travere reserves the right to decline or recommend modifications to a request if it does not comply with the data sharing policy or if it is determined that the request is made by a biased source.
Time Frame: Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication
Access Criteria: Requires submission and approval of intended use and a data sharing agreement.
URL: http://datarequest@travere.com

REFERENCES:
- See also: Sponsor Website — http://travere.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-eight participants were enrolled in the study and all 48 (100%) received at least 1 dose of sparsentan.
  Sparsentan was prematurely discontinued in 9 participants (19%).
  Forty-one participants (85%) completed the study, and 7 participants (15%) discontinued the study. The most common reasons for discontinuation from the study were withdrawal by participant (3 participants [6%]) and AEs (2 participants [4%]).
Pre-assignment Details: 93 participants were screened; 45 participants were screen failures.
  * 29 participants did not meet the inclusion criteria of UA/C ≥0.3 g/g
  * 7 participants did not meet the inclusion criteria of being on a stable dose of ACEI and/or ARB
  * 5 participants did not meet the inclusion criteria of being on a stable dose of an SGLT2 inhibitor
  * 4 participants were excluded for other reasons
Period: Overall Study
Arm/Group | Sparsentan
Started | 48
Discontinued | 7
Completed | 41 (Date of last participant visit.)
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sparsentan
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 48 [19 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 28
  Race: Black or African American | 1
  Race: Asian | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 5
  Ethnicity: Not Hispanic or Latino | 42
  Ethnicity: Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Hong Kong | 11
  United States | 37
Height [Mean (Standard Deviation); unit: centimeters] | 168.2 (11.16)
Weight [Mean (Standard Deviation); unit: Kilograms] | 85.9 (22.25)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.02 (5.619)
Estimated Glomerular Filtration Rate (eGFR) [Number; unit: participants]
  <25 mL/min/1.73m^2 | 0
  >/=25 to <60 mL/min/173m^2 | 33
  >/=60 mL/min/1.73m^2 | 15
Urine protein/creatinine ratio (UP/C) [Geometric Mean (Full Range); unit: g/g] | 1.29 [0.3 to 6.4]
Urine albumin/creatinine ratio (UA/C) [Geometric Mean (Full Range); unit: g/g] | 0.75 [0.2 to 4.1]

OUTCOME MEASURES:

1. Primary Outcome: Change in Urine Albumin-creatinine Ratio (UA/C) at Week 24
Description: The change from baseline in UA/C at Week 24 based on first morning void (FMV) samples
Time Frame: Week 24
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sparsentan
Number analyzed (Participants) | 39
percent change | -55.78 [-65.8 to -42.8]

2. Secondary Outcome: UA/C <0.2 g/g at Week 24
Description: Achievement of UA/C of <0.2 g/g at Week 24 based on FMV samples
Time Frame: Week 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sparsentan
Number analyzed (Participants) | 39
percentage of participants | 31 [17.0 to 47.6]

3. Secondary Outcome: 30% Reduction From Baseline in UA/C at Week 24
Description: Achievement of 30% reduction from baseline in UA/C at Week 24 based on FMV samples
Time Frame: Week 24
Population: UA/C Responder Endpoints While on Treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sparsentan
Number analyzed (Participants) | 39
percentage of participants | 77 [60.7 to 88.9]

4. Secondary Outcome: 50% Reduction From Baseline in UA/C at Week 24
Description: Achievement of 50% reduction from baseline in UA/C at Week 24 based on FMV samples
Time Frame: Week 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sparsentan
Number analyzed (Participants) | 39
percentage of participants | 51 [34.8 to 67.6]

5. Secondary Outcome: Change in Urine Protein-to-creatinine Ratio (UP/C) at Week 24
Description: The change from baseline in UP/C at Week 24 based on FMV samples
Time Frame: Week 24
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Sparsentan
Number analyzed (Participants) | 39
percentage change | -45.20 [-54.6 to -33.9]

6. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: Change from baseline estimated glomerular filtration rate at 24 weeks
Time Frame: Week 24
Population: Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min/1.73 square meter
Arm/Group | Sparsentan
Number analyzed (Participants) | 39
mL/min/1.73 square meter | -2.0 [-3.9 to -0.1]

7. Secondary Outcome: Systolic Blood Pressure (BP) at Week 24
Description: The change from baseline in systolic BP at Week 24
Time Frame: Week 24
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Sparsentan
Number analyzed (Participants) | 39
mmHg | -3.4 [-6.8 to 0.0]

8. Secondary Outcome: Change in Diastolic Blood Pressure (BP)
Description: The change from baseline in diastolic BP at Week 24
Time Frame: Week 24
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Sparsentan
Number analyzed (Participants) | 39
mmHg | -4.6 [-6.7 to -2.4]

ADVERSE EVENTS:
Time Frame: 525 Days (1 year, 5 months, and 6 days) Continuous monitoring from Day -42 (screening) to Week 28 (safety follow-up visit)
Arm/Group | Sparsentan
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 4/48
Other Adverse Events (participants affected / at risk) | 26/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sparsentan (N=48)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular event (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Chemical burn (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sparsentan (N=48)
Hypotension (Vascular disorders) | 7
Headache (Nervous system disorders) | 4
Oedema (General disorders) | 4
Oedema peripheral (General disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Dizziness (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT05856760/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT05856760/SAP_001.pdf